CLINICAL TRIAL: NCT06699524
Title: Construction of a Recurrence Risk Prediction Model for Liver Resection Based on Drug Sensitivity of Patient-derived Liver Cancer Organoid
Brief Title: Construction of a Recurrence Risk Prediction Model for Liver Resection Based on Drug Sensitivity of Patient-derived Hepatocellular Carcinoma Organoid
Status: Active, not recruiting | Type: Observational
Sponsor: Shen Feng (Other)
Responsible Party: Sponsor-Investigator, Shen Feng, Dean of Clinical Research Institute, Director of Four Departments of Hepatology, Chief Physician, Professor, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Other Study IDs: EHBH-202408
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- drug-sensitive group: Organoid resistance and sensitivity are indicated by an IC50 value ≥23.815 μmol/L and < 23.815 μmol/L, respectively. According to the PDTO drug testing, 42 patients were classified into the drug-sensitive group, and 80 patients into the drug-resistant group。
  Interventions: Drug: in vitro （chemotherapy）; Device: Adjuvant TACE（Adjuvant Transarterial Chemoembolization）
- drug-resistant group: Organoid resistance and sensitivity are indicated by an IC50 value ≥23.815 μmol/L and < 23.815 μmol/L, respectively. According to the PDTO drug testing, 42 patients were classified into the drug-sensitive group, and 80 patients into the drug-resistant group。
  Interventions: Drug: in vitro （chemotherapy）; Device: Adjuvant TACE（Adjuvant Transarterial Chemoembolization）

INTERVENTIONS:
Drug: in vitro （chemotherapy） — resuscitating PDTO from the organoid biobank, patients were categorized into drug-sensitive and drug-resistant groups based on the optimal cutoff value for PDTO drug testing. We then followed up to analyze the correlation between PDTO drug testing and RFS.
Device: Adjuvant TACE（Adjuvant Transarterial Chemoembolization） — Adjuvant TACE was performed 4 to 8 weeks postoperatively, with a chemotherapy regimen of 50 mg of doxorubicin and 50 mg of oxaliplatin.

SUMMARY:
Liver cancer is the sixth most common malignant tumor worldwide and the third leading cause of cancer-related deaths. China is a high-risk area for liver cancer, accounting for approximately 55% of primary liver cancer worldwide. Liver cancer is highly malignant and easy to recur, which seriously endangers the life and health of our people. Hepatectomy is the preferred treatment for liver cancer, but the 5-year recurrence rate remains as high as 70%, severely limiting the effectiveness of the surgery. Therefore, exploring the risk factors and predictive methods for early tumor recurrence after liver resection in patients has high clinical value. Clinical practice has found that primary liver cancer patients can be treated with postoperative adjuvant transarterial chemoembolization (TACE) to prevent recurrence. However, the effectiveness of TACE varies among patients and may be related to tumor heterogeneity. However, many studies have reported that drug sensitivity testing based on patient derived organoids can indicate the clinical efficacy of drugs, but there is currently no relevant research indicating that organoids can reflect the therapeutic response of TACE. Therefore, the aim of this study is to explore the correlation between patient derived organoid drug sensitivity testing results and TACE treatment responsiveness and tumor recurrence, and further construct a column chart model to predict tumor recurrence after adjuvant TACE.

ELIGIBILITY:
The inclusion criteria were as follows: (1) age between 18 and 80 years; (2) postoperative pathological diagnosis of HCC; (3) adjuvant TACE performed 4-8 weeks after radical surgical resection; and (4) successful culture of PDTO, with sufficient quantity for drug testing.

The exclusion criteria were as follows: (1) patients with an American Society of Anesthesiologists (ASA) score greater than 3; (2) failure or contamination of PDTO culture; (3) failure to complete standardized adjuvant TACE treatment postoperatively; and (4) patients who received neoadjuvant or other adjuvant therapies, including radiotherapy and systemic treatments.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included samples collected from the organoid biobank of the Eastern Hepatobiliary Surgery Hospital between September 2019 and September 2022.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | Follow-up was performed at least every 2 months during the first 6 months after adjuvant TACE, and every 3 months for the subsequent 18 months. The follow-up period ended in September 2024
  Recurrence within two years post-surgery was classified as early recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Naval Medical University,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided